CLINICAL TRIAL: NCT04173832
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Clinical Study of Treatment of L-DOPA-Induced Dyskinesia With Tianqi Pingchan Granule Combined With Amantadine
Brief Title: Clinical Study on Treatment of L-DOPA-Induced Dyskinesia With Tianqi Pingchan Granule Combined With Amantadine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai University of Traditional Chinese Medicine (Other); Shanghai Municipal Hospital of Traditional Chinese Medicine (Other); Wenzhou Central Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Affiliated Hospital of Nanjing University of Chinese Medicine (Other); The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XHEC-C-2019-032-2
Record Dates: First submitted 2019-10-30; First posted 2019-11-22 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-10

CONDITIONS: L-DOPA-Induced Dyskinesia
MeSH Terms: interventions — Amantadine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tianqi Pingchan Granule Combined With Amantadine (Experimental)
  Interventions: Drug: Tianqi Pingchan Granule Combined With Amantadine
- placebo Combined With Amantadine (Placebo Comparator)
  Interventions: Drug: Placebo Combined With Amantadine

INTERVENTIONS:
Drug: Tianqi Pingchan Granule Combined With Amantadine — Tianqi Pingchan Granule and Amantadine are given to patients simultaneously
  Arms: Tianqi Pingchan Granule Combined With Amantadine
Drug: Placebo Combined With Amantadine — Placebo and Amantadine are given to patients simultaneously
  Arms: placebo Combined With Amantadine

SUMMARY:
A randomized, double-blind, placebo-controlled, multi-center clinical trial was conducted to observe the improvement in the level of dyskinesia in patients with Parkinson's disease during the 12-week period of oral treatment with Tianqi Pingchan Granule Combined With Amantadine. To observe the differences of the safety and effectiveness between Tianqi Pingchan Granule combined with amantadine and placebo combined with amantadine.

ELIGIBILITY:
Inclusion Criteria:

1. PD patients between the ages of 30-85;
2. Patients with Parkinson's disease dyskinesia, and UPDRS 4.2 score ≥ 2 points;
3. The patient diary shows that there are at least two opening periods between 9 am and 4 pm every day, and the dyskinesia appears in the opening period, each time lasting more than half an hour;
4. The treatment plan for anti-Parkinson's disease is stable and not adjusted within 30 days before enrollment;
5. Levodopa is administered at least three times a day.

Exclusion Criteria:

1. PD patients with biphasic, dystonia, closure, myoclonus, but no dyskinesia;
2. pregnant and lactating women;
3. Taking other Chinese medicines against Parkinson's disease 2 weeks before enrollment;
4. Impaired cognitive function (according to pre-entry MMSE score): secondary education level: MMSE <24 points; primary education level <20 points; illiterate <17 points;
5. Psychiatric symptoms associated with anti-Parkinson's disease drugs
6. accompanied by a history of mental illness;
7. impaired liver and kidney function;
8. accompanied by severe other systemic diseases;
9. Amantadine treatment has been received within the first 30 days of enrollment;
10. History of medication with apomorphine or dopamine receptor antagonists;
11. Previously taking amantadine, unable to tolerate;
12. Allergic to the amantadine, memantine, and traditional Chinese medicine preparations or serious adverse reactions;
13. Before the enrollment, the EKG showed obvious abnormalities and required clinical intervention.
14. has received PD-related brain surgery;
15. Patients who are participating in other clinical studies or have participated in other clinical studies within the previous 30 days;
16. Patients who are unable to follow up with follow-up.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Unified Dyskinesia Rating Scale (UDysRS) | up to 12 weeks
  The change from baseline to day 84 of treatment in the sum of the items comprising the Unified Dyskinesia Rating Scale (UDysRS). The UDysRS is administered to assess dyskinesia. The scoring range is 0-104, where higher score means more dyskinesia.

SECONDARY OUTCOMES:
Patient diaries | up to 12 weeks
  Change in daily "OFF"-time as assessed with patient diaries from run-in to day 84. This is a self administered diary where patients assess their motor state every half hour during 24 hours.
Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | up to 12 weeks
  Change in Unified Parkinson's Disease Rating Scale (MDS-UPDRS) total score of part III from Baseline (Day 1) to day 84. The part III of the MDS-UPDRS assess motor function in best on phase. The score range is 0-132, where a higher score means more severe motor impairment.
Clinical Global Impression | up to 12 weeks
  Change score is an ordinal measure of change with a range of 0 (not assessed) to 7 (very much worse). A score of 4 is associated with "no change

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Zhu XB, Zhao Y, Cui GY, Li WT, Yuan CX, Huang JP, Wan Y, Wu N, Song L, Zhao JH, Liang Y, Xu CY, Liu MJ, Gao C, Chen XX, Liu ZG. Efficacy and safety of Tianqi Pingchan Granule, a compound Chinese herbal medicine, for levodopa-induced dyskinesia in Parkinson's disease: A randomized double-blind placebo-controlled trial. J Integr Med. 2024 Sep;22(5):545-551. doi: 10.1016/j.joim.2024.07.002. Epub 2024 Jul 9. PMID 39060125